CLINICAL TRIAL: NCT06774612
Title: Diagnostic Reasoning With and Without AI Support: A Randomized Controlled Trial of LLM-Trained Medical Doctors
Brief Title: The Impact of Large Language Models on Diagnostic Reasoning Among LLM-Trained Medical Doctors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Management Sciences (Other)
Collaborators: King Edward Medical University (Other)
Responsible Party: Principal Investigator, Ihsan Ayyub Qazi, PhD, Associate Professor, PhD, Lahore University of Management Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-0342
Record Dates: First submitted 2025-01-04; First posted 2025-01-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Diagnosis
Keywords: clinical reasoning; large language models; computer-assisted diagnosis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: The trial will be designed as a randomized, two-arm, single-blind parallel group study.
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ChatGPT-4o (Active Comparator): Group will be given access to ChatGPT-4o.
  Interventions: Other: ChatGPT-4o
- Conventional resources (No Intervention): Group will not be given access to ChatGPT-4o but will be encouraged to use any resources they wish besides large language models (PubMed, Google without AI Overviews, etc).

INTERVENTIONS:
Other: ChatGPT-4o — OpenAI's ChatGPT-4o large language model with chat interface.
  Arms: ChatGPT-4o

SUMMARY:
This study aims to evaluate whether large language model-trained medical doctors demonstrate enhanced diagnostic reasoning performance when utilizing ChatGPT-4o alongside conventional resources compared to using conventional resources alone.

DETAILED DESCRIPTION:
Diagnostic errors are a major source of preventable patient harm. Recent advances in Large Language Models (LLM), particularly ChatGPT-4o, have shown promise in enhancing medical decision-making. However, little is known about their impact on medical doctors' (e.g., physicians' and surgeons') diagnostic reasoning.

Diagnostic accuracy relies on complex clinical reasoning and careful evaluation of patient data. While AI assistance could potentially reduce errors and improve efficiency, ChatGPT-4o lacks medical validation and could introduce new risks through incorrect information generation (also known as hallucinations). To mitigate these risks, doctors need adequate training in understanding ChatGPT-4o's capabilities, limitations, and proper usage. Given these uncertainties and the importance of proper AI training, systematic evaluation is essential before clinical implementation.

This randomized study will assess whether ChatGPT-4o access improves LLM-trained medical doctors' diagnostic performance compared to conventional resources (e.g., textbooks, online medical databases) alone. All participating doctors will have completed at least a 10-hour training program covering ChatGPT-4o usage, prompt engineering techniques, and output evaluation strategies. Participants will provide differential diagnoses with supporting evidence and recommended next steps for clinical cases, with responses evaluated by blinded reviewers.

ELIGIBILITY:
Inclusion Criteria:

* Full or Provisionally Registered Medical Practitioners with the Pakistan Medical and Dental Council (PMDC).
* Completed Bachelor of Medicine, Bachelor of Surgery (MBBS) Exam. The equivalent degree of MBBS in US and Canada is called Doctor of Medicine (MD).
* Participants must have completed a structured training program on the use of ChatGPT (or a comparable large language model), totaling at least 10 hours of instruction. The program must include hands-on practice related to LLM's aspects, specifically prompt engineering and content evaluation.

Exclusion Criteria:

* Any other Registered Medical Practitioners (Full or Provisional) with PMDC (e.g., Professionals with Bachelor of Dental Surgery or BDS).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-05-17 (Actual); Study Completion 2025-05-17 (Actual)

PRIMARY OUTCOMES:
Diagnostic reasoning | Assessed at a single time point for each case, during the scheduled diagnostic reasoning evaluation session, which takes place between 0-4 days after participant enrollment.
  The primary outcome will be the percent correct for each case (range: 0 to 100). For each case, participants will be asked for three top diagnoses, findings from the case that support that diagnosis, and findings from the case that oppose that diagnosis. For each plausible diagnosis, participants will receive 1 point. Findings supporting the diagnosis and findings opposing the diagnosis will also be graded based on correctness, with 1 point for partially correct and 2 points for completely correct responses. Participants will then be asked to name their top diagnosis, earning one point for a reasonable response and two points for the most correct response. Finally participants will be asked to name up to 3 next steps to further evaluate the patient with one point awarded for a partially correct response and two points for a completely correct response. The primary outcome will be compared on the case-level by the randomized groups.

SECONDARY OUTCOMES:
Time Spent on Diagnosis | Assessed at a single time point for each case, during the scheduled diagnostic reasoning evaluation session, which takes place between 0-4 days after participant enrollment.
  We will compare how much time (in seconds) participants spend per case between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Ihsan Ayyub Qazi, PhD, Principal Investigator — Lahore University of Management Sciences; Muhammad Asadullah Khawaja, MBBS, Principal Investigator — King Edward Medical University; Ayesha Ali, PhD, Principal Investigator — Lahore University of Management Sciences
Locations (1):
- Lahore University of Management Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No